CLINICAL TRIAL: NCT06282367
Title: Novel Regimen for Colonoscopy Bowel Preparation With Oral Lactulose: A Prospective Comparative Study
Brief Title: Bowel Preparation for Colonoscopy With Oral Lactulose
Status: Completed | Type: Observational
Sponsor: Josue Aliaga (Other Government)
Responsible Party: Sponsor-Investigator, Josue Aliaga, Gastroenterologist, Hospital Jose Agurto Tello
Organization: Hospital Jose Agurto Tello (Other Government)
Other Study IDs: JOSE AGURTO TELLO HOSPITAL
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Colonoscopy; Colonoscopy Preparation
Keywords: bowel preparation; oral lactulose; colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Bowel preparation for colonoscopy using Polyethylene glycol
- Bowel preparation for colonoscopy using oral Lactulose

SUMMARY:
Background and Aims: The quality of colonoscopy is critically influenced by bowel preparation. Polyethylene glycol (PEG) is considered the gold standard regimen for bowel preparation, however due to the necessity of large volume of patient's tolerance is impaired, especially in the elderly population. Lactulose has been adopted in a few centers as a novel alternative for colonoscopy preparation. This study aimed to investigate the efficacy-safety profile of a lactulose-based bowel preparation in comparison to PEG for colonoscopy.

Methods: Prospective non-blinded comparative study, developed in two tertiary centers from July 2021 to April 2023. Outpatients undergoing colonoscopy were randomly divided into 2 groups: Group 1 (111 patients): PEG and Group 2 (111 patients): Lactulose. The following clinical outcomes were assessed for each group: degree of bowel clearance using the Boston Score, colorectal polyp detection rate, adenoma detection rate, tolerability and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ 18 years
* Colorectal cancer screening
* Lower gastrointestinal bleeding
* Iron deficiency anemia
* Chronic diarrhea

Exclusion Criteria:

* Patients with previous colorectal surgery
* Pregnant
* Emergency colonoscopies
* Use of any other scheme or substance for bowel preparation different from those studied
* Incomplete information
* Clinical conditions considered unsuitable for sedation or colonoscopy

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Data were extracted from a prospectively generated database, including consecutive outpatients from July 2021 to April 2023 who underwent diagnostic colonoscopy
Sampling Method: Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Degree of bowel cleansing using the Boston score | 21 month
  minimum value: 0 (worse outcome: inadequate bowel preparation); maximum value: 9 (better outcome: adequate bowel preparation)

SECONDARY OUTCOMES:
adenomas detection rate | 21 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jose Agurto Tello Hospital, Lima, Peru